CLINICAL TRIAL: NCT06627296
Title: The Effect of Combined Exercise Training With Neuromuscular Electrical Stimulation on Muscle Strength, Proprioceptive Sense, Reaction Time, and Functionality in Patients Diagnosed With Scapholunate Instability
Brief Title: The Effect of Combined Exercise and NMES on Strength, Proprioception and Reaction Time in Scapholunate Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Arzu Dağ, Doctorate student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/626
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Scapholunate Interosseous Ligament Injury; Scapholunate Dissociation; Scaphoid-Lunate Instability
Keywords: Scapholunate Instability; Neuromuscular Electrical Stimulation; Isokinetic Muscle Strength; Proprioceptive Sensation; Reaction Time; Functionality
MeSH Terms: interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups with a intervention group including Nmes and exercise therapy and a control group including exercise therapy
Who Masked: Outcomes Assessor
Masking Description: Blinding was done by ensuring that the participant did not know which group the subject was they were in. Also, the other researcher assessing the measurements did not know which treatment the patients received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation Group combined with Exercise Training (Experimental): The intervention group will receive neuromuscular electrical stimulation combined with exercise training. The group will also be given home exercises to continue at home.
  Individuals in the NMES group will undergo NMES application accompanied by a physiotherapist for a total of 24 sessions of 15 repetitions 3 days a week for 8 weeks and then exercise programs will be performed face-to-face.
  On the other days, patients will be asked to perform 3 sets of 15 repetitions every day as home exercises.
  Exercise training includes intrinsic and extrinsic muscle strengthening, wrist stabilization exercises, dart exercises, wrist neuromuscular exercises using different materials, reactive muscle control, perturbation exercises.
  Interventions: Other: Exercise Training; Device: Neuromuscular Electrical Stimulation
- Exercise Training Group (Control Group) (Experimental): Patients in the control group will have face-to-face exercise programs with a physiotherapist. Exercise training includes intrinsic and extrinsic muscle strengthening, wrist stabilization exercises, dart exercises, wrist neuromuscular exercises using different materials, reactive muscle control, perturbation exercises.
  Interventions: Other: Exercise Training (Control Group)

INTERVENTIONS:
Other: Exercise Training — Individuals in the NMES group will have a total of 24 sessions of NMES application with 15 repetitions 3 days a week for 8 weeks and then exercise programs will be performed face-to-face. They will also be given home exercises to continue at home.
  In the NMES group, NMES training will be performed for extensor carpi radialis longus (ECRL), extensor carpi radialis brevis (ECRB), abductor pollicis longus (APL), flexor carpi radialis (FCR) muscles. The pencil electrode will be used to stimulate the ECRL, ECRB, FCR and APL muscles in such a way that 30+30+30=90 contractions will be obtained from each muscle. According to the morphologic characteristics of each muscle, different current and will be applied.
  P11th program to ECRL and APL : 65 Hz. 200 μs, P13th program to ECRB and FCR 50 Hz, 200 μs will be applied. Exercises includes intrinsic and extrinsic muscle strengthening, stabilization exercises and dart exercises, wrist neuromuscular exercises and perturbation exercises.
  Arms: Neuromuscular Electrical Stimulation Group combined with Exercise Training
Other: Exercise Training (Control Group) — Patients in the control group will have face-to-face exercise programs with a physiotherapist for a total of 24 sessions of 15 repetitions 3 days a week for 8 weeks. Exercises will be performed 3 days a week with a physiotherapist. On the other days, patients will be asked to perform 3 sets of 15 repetitions every day as home exercises.
  Exercise training includes intrinsic and extrinsic muscle strengthening, wrist stabilization exercises, dart exercises, wrist neuromuscular exercises using different materials, reactive muscle control, perturbation exercises.
  Exercises will be at the limit of pain. Until the 6th month, overloading, strong gripping, weight transfer, rotations and lifting heavy objects should be avoided. Rehabilitation with functional range of motion is important. Exercises will be performed with a physiotherapist 3 days a week. On the other days, patients will be asked to perform 3 sets of 15 repetitions every day as home exercises.
  Arms: Exercise Training Group (Control Group)
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation
  Arms: Neuromuscular Electrical Stimulation Group combined with Exercise Training

SUMMARY:
In our study, which we conducted to investigate the effect of exercise training combined with neuromuscular electrical stimulation on muscle strength, proprioceptive sensation, reaction time and functionality in patients with scapholunate (SL) instability, individuals with SL instability who meet the inclusion criteria and volunteer to participate in the study will participate. After the approval of the ethics committee, it is planned to include as many individuals with SL instability as the number to be obtained following the power analysis to be performed as a result of the pilot study. The pain of the subjects will be evaluated with the VAS pain scale during rest-activity-exercise. All participants will be evaluated with the isokinetic cybex device for isokinetic muscle strength of the wrist, grip strength with the JAMAR hand held dynometer, NEH evaluation: goniometer, proprioceptive sensation with ACUMAR and isokinetic device, reaction time with blazepod trainer, wrist pain transfer with a digital scale, assessment of upper extremity functional status: pwre (patient rated wrist evaluation), modified mayo wrist score, DASH, EL20 questionnaire, SF-12 questionnaires.

In this randomized controlled study, the first group will receive NMES and exercise training 3 days a week for a total of 8 weeks and the other group will receive only exercise training. The evaluations will be done at the beginning and twice in total after the 8-week rehabilitation program. The exercises given to the patients in both groups will be similar for 8 weeks and they will receive a total of 24 sessions of exercise programs with 15 repetitions per day, 3 days a week, accompanied by a physiotherapist. Both groups will also be given home exercises to continue at home. NMES and exercise trainings will be applied in such a way that activation of SL-friendly extensor carpi radialis longus (ECRL), extensor carpi radialis brevis (ECRB), flexor carpi radialis (FCR), and abductor pollicis longus (APL) muscles will be followed by inhibition of non-friendly extensor carpi ulnaris (ECU).

After the completion of the thesis, it is planned to add to the literature by examining the effects of exercise training combined with NMES on muscle strength, proprioceptive sensation, reaction time and functionality in individuals diagnosed with SL instability and the superiorities, if any, between the methods.

DETAILED DESCRIPTION:
Among upper extremity injuries, hand/wrist injuries are frequently observed. The hand is an important organ that enables individuals to perform daily life activities. Hand and wrist problems can cause limitations in the person's activities and prevent the person from fulfilling daily life roles. This can lead to a decrease in quality of life.

n terms of biomechanical properties, extrinsic ligaments of wrist show greater elasticity but are less resistant to traction, resulting in lower durability compared to most intrinsic ligaments. As a result, extrinsic ligaments are prone to rupture in the medial portions, whereas intrinsic ligaments are more prone to rupture injuries rather than a complete tear (1).

The scapholunate (SL) joint relationship is provided by several carpal ligaments. The most important of these is the scapholunate interosseous ligament (SLIL; scapholunate interosseous ligament) (2). SLIL injury results in scapholunate joint instability (3). Scapholunate instability is the most common carpal instability (4). When this instability is left untreated, the mechanical relationship between the carpal bones is permanently disrupted, resulting in progressive degenerative changes in the radiocarpal and midcarpal joints (5). These degenerative changes are called scapholunate advanced collapse (SLAC) and are the most common cause of wrist osteoarthritis (6). In SL instability, extension and falling on the hand in ulnar deviation typically constitute the mechanism of injury. The combined pattern of carpal instability and degenerative arthritis is called scapholunate advanced collapse (SLAC) (7).

The fact that the scaphoid and lunate have different articular structures allows them to rotate at different rates during wrist flexion and extension movements. In addition, the dorsal fibers of the SLIL are short and thick and the palmar fibers are loose and elastic, allowing different rotations of the scaphoid and lunate during flexion and extension movements. With loading, the scaphoid tends to go into flexion and the lunate tends to go into extension. These different movement patterns of the scaphoid and lunate result in a high potential energy stored in the SLIL ligament. When ligament rupture occurs, the carpal bones are expected to move to the opposite side due to this energy. Therefore, after SLIL rupture, the scaphoid flexes and the lunate goes into extension due to the pulling effect of the triquetrum through the lunatriquetral interosseal ligament (LTIL). This instability pattern is called dorsal intercalary segment instability (DISI) (7).

Until recently, most biomechanical theories suggested that wrist stability was mainly determined by the shape of the joint and the interaction between ligaments and capsules. The dynamic stabilization mechanisms of other joints such as the knee or shoulder have been extensively investigated. Less emphasis has been placed on understanding how muscles and tendons contribute to wrist stability. However, over the last 15 years, increasing interest and research has started to shed light on this topic. In fact, more than 350 articles on wrist proprioception have been published since 2011. One of the triggers for this fact was the description of mechanoreceptors in the wrist ligaments by Hagert et al. Proprioception is related to joint stability. The term "wrist stability" refers to the ability of the wrist to maintain balance under load (kinetic) and/or during movement (kinematic), and can persist strongly without twisting and becoming symptomatic. A stable wrist does not twist under physiological load and can adjust its internal alignment to become a solid block from which forces can be distributed. Kinetic stability of the wrist requires many contributing factors, including bone morphology, robust static (ligaments) and strong dynamic stabilizers (forearm muscles and tendons crossing the wrist), preserved articulating surfaces, and a competent sensory and motor system that includes nerves connecting the static and dynamic stabilizers. Failure of any of these five factors can lead to wrist instability (13).

SL instability occurs as a result of disruption of the normal alignment of the bones forming the wrist due to damage to the SLIL ligaments. It is often overlooked because it may be associated with other hand/wrist problems (14,15). SL instabilities are usually characterized by wrist pain that occurs during loading. The pain pattern developing due to SL instability increases during activity. Pain may lead to loss of normal joint movements and decreased grip strength. This leads to incompetence in activities of daily living and self-care and a decrease in functional level (16-18). Different factors are considered in the treatment of SL instability problems.

In recent years, studies on carpal kinetics, kinematics and ligament properties have shed light on conservative treatment approaches (21-23). Different rehabilitation approaches have been developed especially by investigating the ligaments and muscles that contribute to carpal stability (24,25). In a study by Hagert et al. (26), it was reported that one of the most important factors contributing to carpal stability is proprioceptive and neuromuscular control of the wrist joint. In their study investigating the structural and neural properties of the wrist ligaments, they noted that the ligaments adhering to the dorsal and tricuetrum, especially the scapholunate interosseous ligament (SLIL), were rich in mechanoreceptors (27). In addition, the presence of ligamentomuscular reflexes that cause activity in the forearm muscles as a result of electrical stimulation of the SLIL has been demonstrated.

It has been shown that especially the flexor carpi ulnaris (FCU), flexor carpi radialis (FCR), extensor carpi radialis longus (ECRL), extensor carpi ulnaris (ECU) and extensor carpi radialis brevis (ECRB) muscles play an effective role in dynamic stabilization of the wrist. In a study by Garcia-Ellias et al. (29), it was shown that these muscles change the distance between the carpal bones by making the carpal bones pronate or supinate. As a result of these studies, the idea that further injuries can be prevented by activating the right muscles after ligament damage has emerged (29).

In their study on cadavers, Salva-Coll et al. investigated the movement patterns of the FCU, FCR, ECRL, ECU and Abductor Pollicis Longus (APL) muscles on the carpal bones. It was noted that the FCU, ECRL and APL muscles caused supination of both carpal rows, especially flexion of the proximal carpal row (30). It has been observed that the FCR muscle supinates the scaphoideum and pronates the tricuetrum and capitatum. The ECU muscle was found to pronate both the distal and proximal carpal row significantly (31). It was noted that carpal supination narrowed the scapholunate interval, while pronation widened it. Therefore, the ECRL, APL, and FCR muscles, which are defined as "scapholunate friendly" after SLL injuries, have gained importance in the rehabilitation of carpal instability because they narrow the scapholunate space (32). It has also been reported that ECU activity should be avoided.

Studies have reported that simultaneous excitation of the ECR, FCR and FCU and their muscles can provide global stability of the wrist joint. Therefore, co-activation exercises are recommended to be included in the rehabilitation program to increase dynamic stability (7) Electrical stimulation is widely used for skeletal muscle strengthening.

Neuromuscular electrical stimulation (NMES) is a method that reorganizes the central nervous system, causes biochemical, physiological and histological changes in muscle fibers, prevents muscle atrophy and facilitates the recovery of muscle strength and function in patients with central nervous system lesions (33). Studies have shown that NMES applied to the unilateral extremity provides an increase in muscle strength (34).

In the literature, it has been reported that NMES causes an increase in the pennation angle and physiological cross-sectional area (PCSA) values of muscles as a result of some physiologic processes (35,36). Especially currents below 50 Hz are suitable for muscles with short fiber length and high PCSA values because they contain long durations. In other words, low frequency long duration selections will be appropriate for pennate muscles. For muscles with low PCSA and high fiber length values, the selection parameters will be different. For these muscles, frequencies above 70 Hz and very short (approximately 200 µsec) durations should be preferred and stimulation times should be kept short (35-37).

Shardong et al. (38) showed that muscle strength increased after eight weeks of NMES intervention in patients with chronic renal failure, but muscle 2 thickness and pennation angle did not change. Variable NMES parameters (frequency, amplitude, duration, electrode placement, etc.) have been shown as the reason for these conflicting results regarding the effects of NMES (39).

In the current literature published by Salva-Coll et al. in 2023, it is thought that there may be an imbalance of flexor and extensor muscles of the forearm muscles due to damage to the ligamentomuscular reflex mechanism arising from the SLL after SLL injury. It has been reported that the above-mentioned ECRL, ECRB, APL, FCR muscles are important in the rehabilitation of carpal instability because they narrow the scapholunate space and ECU activity should be avoided. In case reports, it is described that neuromuscular rehabilitation of dynamic stabilizers of this wrist, which is thought to be "SL joint friendly", is applied. The use of an arc of motion called the dart throwing motion has also become widespread in rehabilitation. It has been shown to minimize the load on the SLIL and is a widely used application in postoperative SLIL rehabilitation (40). These approaches have been derived from basic science literature, rehabilitation concepts available for other anatomical locations, and biomechanical investigations of the wrist. However, there is limited evidence to explain the effectiveness of these practices. There are no randomized clinical trials or guidelines in the literature that recommend ideal conservative rehabilitation strategies for SLIL injuries. Given the paucity of literature, it is still inevitable that rehabilitation clinicians intervene in patients with SLIL injuries.

The effect of NMES on isokinetic muscle strength, grip strength, joint proprioception in scapholunate patients is unknown in the literature. It is important to understand the effect of NMES on the muscles mentioned above as SL joint friendly in order to achieve a more effective treatment outcome in patients.

There are no studies in the literature that apply NMES to SL friendly muscles in patients with SL instability. In the existing studies, there are studies that include general wrist exercise training after surgery. Among these studies, there were no studies investigating wrist extensor and flexor isokinetic muscle strength and endurance after exercise training. In addition, in the existing studies, randomized controlled studies measuring upper extremity reaction time, proprioceptive sensation and wrist pain transfer power were not found in SL patients after injury. However, proprioceptive sensation, reaction speed and reaction time are very important for upper extremity functionality. In addition, it is obvious that having an idea about the muscle strength of extensors and flexors with isokinetic measurements will shape rehabilitation protocols differently.

In this study, we aimed to investigate the effect of exercise training combined with neuromuscular electrical stimulation on muscle strength, proprioceptive sensation, reaction time and functionality in patients with scapholunate instability.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Applying to the clinic within the last 6 months
* Being diagnosed with scapholunate instability

Exclusion Criteria:

* Having a history of previous hand/wrist surgery
* Having a neurological or severe systemic disease
* Having any entrapment neuropathy in the upper extremity
* Having any trauma in the upper extremity
* Having a history of reflex sympathetic dystrophy
* Being diagnosed with cervical disc herniation
* Having a psychiatric disorder that will affect cooperation
* Having received training focused on sensory and functional rehabilitation in either hand in the last 6 months
* For any reason, the patient and family do not want to participate in the study or do not comply with the tests.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-08-09 (Actual)

PRIMARY OUTCOMES:
Hand Isokinetic Muscle Strength Evaluation | 1 day before intervention
  It will be evaluated with the Isokinetic Cybex device. At 60/90/ angular velocities, the extensor-flexor peak torque force / work produced by the muscle will be evaluated concentrically.
Hand Isokinetic Muscle Strength Evaluation | 1 day of discharge
  It will be evaluated with the Isokinetic Cybex device. At 60/90/ angular velocities, the extensor-flexor peak torque force / work produced by the muscle will be evaluated concentrically.
Grip Strength Evaluation | 1 day before intervention
  It will be evaluated with the JAMAR hand held dynamometer
Grip Strength Evaluation | 1 day of discharge
  It will be evaluated with the JAMAR hand held dynamometer
Wrist Proprioception Evaluation | 1 day before intervention
  It will be evaluated with the Isokinetic Cybex Device and ACUMAR device The hand will be brought to the target angle value of 30 degrees extension or 30 degrees flexion with the help of a physiotherapist and will be waited for approximately 5 seconds. After the patient learns, he/she will be asked to do it himself/herself with his/her eyes closed. After the movement is repeated 3 times in a row, the participant will be asked to actively apply the determined target extension movement to the same extremity. The difference between the target angle and the measured angle. The difference between the target angle and the measured angle will be recorded as the margin of error.
Wrist Proprioception Evaluation | 1 day of discharge
  It will be evaluated with the Isokinetic Cybex Device and ACUMAR device The hand will be brought to the target angle value of 30 degrees extension or 30 degrees flexion with the help of a physiotherapist and will be waited for approximately 5 seconds. After the patient learns, he/she will be asked to do it himself/herself with his/her eyes closed. After the movement is repeated 3 times in a row, the participant will be asked to actively apply the determined target extension movement to the same extremity. The difference between the target angle and the measured angle.The difference between the target angle and the measured angle will be recorded as the margin of error.
Pain Evaluation: Visual Analog Scale | 1 day before intervention
  It contains 10 cm line that should be assigned according to perceived pain intensity at rest, during activity and while exercising.
Pain Evaluation: Visual Analog Scale | 1 day of discharge
  It contains 10 cm line that should be assigned according to perceived pain intensity at rest, during activity and while exercising.
Evaluation of Reaction Time | 1 day before intervention
  Upper extremity reaction time evaluation will be performed with the reaction speed measurement and exercise set Blazepod Trainer (Blazepod Trainer Device, Play Coyotta Ltd. Tel Aviv Israel) device. Individuals will be asked to turn off the 5 LEDs placed on the table in front of them as quickly as possible with one hand in the sitting position. Both hands will be evaluated. The number of LEDs extinguished in 30 seconds (number), the unit extinguishing time (msec) and the number of LEDs missed when the LEDs extinguished after a 5-second waiting period will be recorded. Measurements will be made on both hands.
Evaluation of Reaction Time | 1 day of discharge
  Upper extremity reaction time evaluation will be performed with the reaction speed measurement and exercise set Blazepod Trainer (Blazepod Trainer Device, Play Coyotta Ltd. Tel Aviv Israel) device. Individuals will be asked to turn off the 5 LEDs placed on the table in front of them as quickly as possible with one hand in the sitting position. Both hands will be evaluated. The number of LEDs extinguished in 30 seconds (number), the unit extinguishing time (msec) and the number of LEDs missed when the LEDs extinguished after a 5-second waiting period will be recorded. Measurements will be made on both hands.
Weight-Bearing Test | 1 day before intervention
  Test protocol: The subject will be asked to apply as much pressure as possible with the extended elbow and wrist on a digital scale. The subjects will perform 3 trials and the average value will be recorded in kilograms and will be compared with the weight transfer test of the unaffected hand, which is determined as a normative value for maximum weight-bearing capacity.
Weight-Bearing Test | 1 day of discharge
  Test protocol: The subject will be asked to apply as much pressure as possible with the extended elbow and wrist on a digital scale. The subjects will perform 3 trials and the average value will be recorded in kilograms and will be compared with the weight transfer test of the unaffected hand, which is determined as a normative value for maximum weight-bearing capacity.

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation (PWRE) | 1 day before intervention
  PRWE is the Patient-Rated Wrist Evaluation.The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. Developed in 1998 for clinical assessment and is used for specific wrist problems.It is one of the reliable upper extremity outcome instrument
Patient Rated Wrist Evaluation (PWRE) | At the time of discharge
  PRWE is the Patient-Rated Wrist Evaluation.The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. Developed in 1998 for clinical assessment and is used for specific wrist problems.It is one of the reliable upper extremity outcome instrument
Modified Mayo Wrist Score | 1 day before intervention
  he Modified Mayo Wrist Score (MMWS)3 is a modification of the Geen and O'Brien score.4 There is a total of 100 points which are divided among the evaluator's assessment of pain (25 points), active flexion/extension arc as a percentage of the opposite side (25 points), grip strength as a percentage of the opposite side (25 points), and the ability to return to regular employment or activities (25 points). Pain is rated as none (25 points), mild (20 points), moderate (10 points), or severe (0 points) by the evaluator, based on the patient's subjective description. The total score ranges from 0 to 100 points with higher scores indicating a better result. An excellent result is defined as 90-100 points, good is 80-89, fair is 65-79 points, and poor is less than 65 points.
Modified Mayo Wrist Score | At the time of discharge
  he Modified Mayo Wrist Score (MMWS)3 is a modification of the Geen and O'Brien score.4 There is a total of 100 points which are divided among the evaluator's assessment of pain (25 points), active flexion/extension arc as a percentage of the opposite side (25 points), grip strength as a percentage of the opposite side (25 points), and the ability to return to regular employment or activities (25 points). Pain is rated as none (25 points), mild (20 points), moderate (10 points), or severe (0 points) by the evaluator, based on the patient's subjective description. The total score ranges from 0 to 100 points with higher scores indicating a better result. An excellent result is defined as 90-100 points, good is 80-89, fair is 65-79 points, and poor is less than 65 points.
Quick DASH | 1 day before intervention
  The QuickDASH is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Quick DASH | At the time of discharge
  The QuickDASH is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Hand20 Questionnaire | 1 day before intervention
  Hand20 was developed to assess upper extremity disorders. During the process of item selection, Suzuki et al. tried to choose items that appeared to reflect the function of the upper extremities and were the least affected by cultural differences. It is composed of 20 short questions accompanied by explanatory illustrations that elderly people and children can easily understand (19 of the 20 questions).
Hand20 Questionnaire | At the time of discharge
  Hand20 was developed to assess upper extremity disorders. During the process of item selection, Suzuki et al. tried to choose items that appeared to reflect the function of the upper extremities and were the least affected by cultural differences. It is composed of 20 short questions accompanied by explanatory illustrations that elderly people and children can easily understand (19 of the 20 questions).
12-Item Short Form Survey (SF-12) | 1 day before intervention
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study[1]. The SF-12 was created to reduce the burden of response.
12-Item Short Form Survey (SF-12) | At the time of discharge
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study[1]. The SF-12 was created to reduce the burden of response.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Topuz, Prof.Dr., Principal Investigator — Hacettepe University; Arzu Dağ, Ph.D Student, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Physical Therapy and Rehabilitation, Hacettepe University, Ankara, Sıhhiye Campus Hacettepe University Sıhhiye, Ankara
  - İstanbul University İstanbul Faculty of Medicine, Istanbul, Çapa, Fatih

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dag A, Ayik O, Firat T, Sahinkaya T, Topuz S. The effectiveness of NMES-integrated therapy in scapholunate ligament injuries - a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Dec 2;18(1):12. doi: 10.1186/s13102-025-01452-4. PMID 41331647